CLINICAL TRIAL: NCT05779085
Title: ASSESSMENT OF CLINICAL, INSTRUMENTAL AND NOTICED EFICACY BY SUBJECTS OF A COSMETIC PRODUCT 12.0417.01.090 UNDER NORMAL CONDITIONS OF USE Study With Dermatological Follow-up Including Instrumental Measurements
Brief Title: Efficacy of a Deep Cleansing Gel Containing 2% Salicylic Acid, 0.2% Zinc Gluconate and 0.05% Lipohydroxy Acid in the Management of Mild to Moderate Facial Acne
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: 090.324.003.12
Record Dates: First submitted 2023-03-07; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Acne Vulgaris on the Face

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dermocosmetic — Use of daily cleanser to treat facial acne
  Other Names: Cleanser

SUMMARY:
A clinical study with 56 healthy subjects (both sexes) aged between 13 to 25 years old. Subjects enrolled had a minimum of 5 inflammatory lesions (papules, nodules and pustules) and 10 non-inflammatory lesions (open and closed comedones), determined by dermatologist. The clinical evaluation considered in oiliness, shininess and global aspect of the skin too. Instrumental assessment of oiliness and shininess was performed, respectively, by Sebumeter and Sebutape.

IThe tested cleanser was used twice daily (morning and evening) during 28 days.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 13-25 years
* mild to moderate acne on the face
* signed informed consent

Exclusion Criteria:

* subjects below 13 years and above 26 years
* severe acne on the face

Ages: 13 Years to 26 Years | Sex: All
Age Groups: Child, Adult
Study Population: Subjects aged between 13 to 25 years of age with mild to moderate acne.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2013-04-08 (Actual); Primary Completion 2013-07-22 (Actual); Study Completion 2013-07-22 (Actual)

PRIMARY OUTCOMES:
Global lesion count | baseline
  using GEA scale
Global lesion count | Day 28
  using GEA scale
Closed comedones | baseline
  count
Closed comedones | Day 28
  count
papules | baseline
  count
papules | Day 28
  count
skin oiliness | baseline
  instrumental measurement Sebumeter
skin oiliness | Day 28
  instrumental measurement Sebumeter
skin sebutape | baseline
  instrumental measurement Sebumeter
skin sebutape | Day 28
  instrumental measurement Sebumeter
subject satisfaction | Day 28
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Carlos Tortely Hospital, Niterói, Brazil

IPD SHARING:
Plan to Share IPD: No